CLINICAL TRIAL: NCT06843681
Title: Trastuzumab Combined With Taxane Neoadjuvant Therapy for HER2-positive Breast Carcinoma in Situ: a Phase II Single-arm Clinical Study
Brief Title: Trastuzumab Plus Taxane Neoadjuvant Therapy for HER2-Positive Breast Ductal Carcinoma In Situ (DCIS) : A Phase II Study
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-746-01
Record Dates: First submitted 2024-12-26; First posted 2025-02-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Carcinoma in Situ
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): The study includes a single treatment arm where all participants will receive a combination of trastuzumab and taxane as part of the neoadjuvant therapy. This treatment arm is designed to assess the efficacy and safety of the regimen in patients with HER2-positive breast carcinoma in situ
  1. Trastuzumab (HER2-Targeted Therapy):
     * Trastuzumab will be administered intravenously at a standard dosage based on the patient's body weight. The initial dose will be a loading dose followed by maintenance doses every three weeks, as per clinical guidelines for HER2-positive breast cancer treatment.
     * The therapy targets the HER2 receptor to inhibit tumor growth and improve response rates.
  2. Taxane (Chemotherapy):
     * A taxane-based chemotherapeutic agent (e.g., paclitaxel or docetaxel) will be administered intravenously. The specific agent, dosage, and schedule will follow standard protocols used in the neoadjuvant setting for HER2-positive breast cancer.
     * Taxanes work by disrupting microt
  Interventions: Drug: Trastuzumab combined with taxane neoadjuvant therapy

INTERVENTIONS:
Drug: Trastuzumab combined with taxane neoadjuvant therapy — Trastuzumab combined with taxane neoadjuvant therapy

SUMMARY:
This is a phase II single-center single-arm clinical study designed to analyze the efficacy and safety of trastuzumab combined with taxane neoadjuvant therapy for HER2-positive breast carcinoma in situ (or with invasive carcinoma).

DETAILED DESCRIPTION:
This Phase II single-center, single-arm clinical study was designed to evaluate the efficacy and safety of trastuzumab combined with taxane as a neoadjuvant treatment for patients with HER2-positive breast cancer in situ or invasive breast cancer. The study was designed to determine breast-conserving surgery rates and pathologic complete response (pCR) rates, assess tumor size reduction, and evaluate potential adverse events associated with treatment options. Participants will be treated with trastuzumab and taxane on a prescribed schedule, with periodic evaluations including imaging, histopathological analysis, and safety monitoring. The aim is to gain insight into the therapeutic potential of this combination therapy in improving outcomes for patients with HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed breast carcinoma in situ (female, 18 to 70 years old);
2. Breast mass ≥2cm, and in situ cancer pathology confirmed HER2 positive (definition: immunohistochemical results 3+ or in situ hybridization results positive);
3. No evidence of distant transfer;
4. Have not received any previous cancer treatment;
5. Imaging examination showed at least one measurable lesion within 2 weeks before enrollment;
6. Left ventricular ejection fraction (LVEF) was measured by echocardiography ≥50%;
7. Previous treatment-related toxicity should be alleviated to NCI CTCAE (version 5.0) ≤1 degree, AST and ALT≤2.5 times the upper limit of normal, total bilirubin ≤1.5 times the upper limit of normal;
8. Liver and kidney function tests are basically normal:

   1. Total bilirubin (TBIL) ≤3× upper limit of normal (ULN),
   2. Alanine aminotransferase and aspartate aminotransferase (ALT/AST) ≤2.5×ULN (patients with liver metastasis ≤5xULN),
   3. Serum creatinine ≤1.5×ULN or creatinine clearance (Ccr) ≥60 ml/min;
9. Adequate bone marrow functional reserve:

   1. White blood cell count (WBC) ≥3.0×10^9 / L,
   2. Neutrophil count (ANC) ≥1.5×10^9 / L,
   3. Platelet count (PLT) ≥70×10^9 / L
10. Fertile women must use contraceptives;
11. Be able to understand the research process, voluntarily participate in the study, and sign the informed consent.

Exclusion Criteria:

1. Metastatic breast cancer (stage IV);
2. History of invasive breast cancer, or prior systemic treatment to treat or prevent breast cancer;
3. Previous or concurrent malignant diseases, except skin basal cell carcinoma or cervical cancer in situ;
4. Patients with severe heart disease or discomfort that is not expected to tolerate chemotherapy, including but not limited to: fatal arrhythmias or higher grade atrioventricular block, unstable angina pectoris, clinically significant valvular disease, transmural myocardial infarction shown by electrocardiogram, uncontrolled hypertension;
5. Insufficient bone marrow or kidney function, liver function impairment;
6. Grade 2 or more severe peripheral neuropathy;
7. Patients with thrombocytopenia, neutropenia, anemia, hypokalemia, and elevation of alanine aminotransferase or aspartate aminotransferase above CTCAE Level 1;
8. Patients who are known to be allergic to the active ingredient or other ingredient of the investigational drug;
9. Had received radiotherapy, chemotherapy, endocrine therapy, or was participating in any interventional drug clinical trial within 4 weeks prior to enrollment;
10. Pregnant or lactating women, women of childbearing age who refused to use effective contraception during the study period;
11. Any other conditions that the investigator considers the patient unfit to participate in the study, concomitant diseases or conditions that may interfere with study participation, or any serious medical disorder that may affect the safety of the subject (e.g., uncontrolled heart disease, high blood pressure, active or uncontrollable infection, active hepatitis B virus infection).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Breast-conserving surgery rate after 4-6 cycles of treatment | From the start of neoadjuvant therapy to the completion of surgery (approximately 3-4 months after enrollment)
  The breast-conserving surgery rate was calculated as a percentage of the total number of patients who successfully completed breast-conserving surgery after neoadjuvant therapy. For this study, all patients were required to confirm after treatment that the tumor was resectable and had no significant metastasis by imaging evaluation, such as breast ultrasound or MRI.

SECONDARY OUTCOMES:
pathological Complete Response (pCR) | Within 3-4 months from enrollment, at the completion of neoadjuvant therapy.
  pCR refers to the situation in which a patient's carcinoma in situ tumor has completely disappeared through pathological examination after neoadjuvant therapy.
  Measurement Tool: Histopathological examination of surgical specimens.
Objective Response Rate (ORR) | Within 3-4 months from enrollment, at the completion of neoadjuvant therapy.
  ORR is the proportion of patients whose tumors have shrunk significantly over the course of treatment. Specifically, ORR includes both partial response (PR) and complete response (CR). Partial response (PR) : The maximum diameter or volume of the tumor is reduced by at least 30%, but it does not completely disappear. Complete response (CR) : The tumor disappears completely and no visible signs of cancer are confirmed by imaging tests, such as CT scans, MRI, or ultrasound.
  Measurement Tool: Imaging assessments (MRI, CT, or ultrasound).
Event-free survival (EFS) of 3 years | At 36 months from the date of enrollment.
  Event-free survival (EFS) is defined as the time from the initiation of neoadjuvant therapy to the first occurrence of disease progression, recurrence, second primary cancer, or death from any cause. In this study, 3-year EFS is defined as the proportion of patients who have not experienced any of these events within 36 months after starting treatment.
  Measurement Tool: Clinical and imaging follow-ups, verified by medical records.
Event-free survival (EFS) of 5 years | At 60 months from the date of enrollment.
  Measurement Tool: Clinical and imaging follow-ups, verified by medical records.
Overall survival | From enrollment to 60 months ± 3 months or until the date of death from any cause, whichever occurs first.
  Measurement Tool: Survival status verified through medical records and patient follow-up.
Biomarker analysis o f HER2 and Ki-67 using immunohistochemistry (IHC) or quantitative PCR | Within 4-6 months from enrollment, at the completion of surgery.
  Measurement Tool: Expression levels of specific biomarkers, such as HER2 and Ki-67, will be assessed using immunohistochemistry (IHC) or quantitative PCR, with tumor tissue or blood samples collected at baseline and post-therapy.
AE rate | From enrollment to 12 months after the end of study treatment.
  Adverse event rate
Assessment of quality of life in patients using the FACT-B scale | From enrollment to 12 months after the end of study treatment or the last follow-up visit.
  Quality of life refers to people's perception and experience of their physical state, mental function, social ability, and overall personal situation based on socioeconomic, cultural background and value orientation. FACT-B scale was used to assess patients before treatment, during treatment (from the first day of the third cycle, and every two cycles thereafter), and 30 days after treatment. Patients' quality of life was quantified by the proportion of changes in the score

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China